CLINICAL TRIAL: NCT01717131
Title: A Non Inferiority Randomized Multicenter Phase III Trial of Axillary Node Dissection Versus no Axillary Node Dissection in Case of Positive Sentinel Lymph Node in Invasive Breast Cancer
Brief Title: Axillary Node Dissection Versus no Dissection in Breast Cancer With Positive Sentinel Lymph Node
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SERC / IPC 2012-001
Record Dates: First submitted 2012-10-19; First posted 2012-10-30 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Invasive Breast Cancer
Keywords: Invasive breast cancer
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery for standard axillary node dissection (Active Comparator): Standard axillary dissection
  Interventions: Procedure: Surgery for standard axillary node dissection
- No axillary lymph node dissection (Experimental): No surgery of axillary lymph node In this study, the absence of surgery is the experimental arm (non-inferiority trial)
  Interventions: Other: No axillary lymph node dissection

INTERVENTIONS:
Procedure: Surgery for standard axillary node dissection
  Arms: Surgery for standard axillary node dissection
Other: No axillary lymph node dissection — No surgery on axillary lymph node
  Arms: No axillary lymph node dissection

SUMMARY:
Data from cohorts, prospective studies and one randomized trial (ASCOG Z0011) support the hypothesis that omission of additional axillary dissection in case of positive sentinel node has a limited impact on overall survival and relapse free survival. However, these data are not sufficient enough to recommend, as a standard of care, to avoid axillary dissection in case of positive sentinel node. The ASCOG Z0011 trial has been closed before the end of inclusions and the predefined non inferiority margin was found to be too large (5% difference at 5 years for primary endpoint).

Prospective randomized trial is then urgently mandatory before omission of axillary node dissection becomes a usual practice without a sufficient scientific level of proof. Indeed, in several reviews, the rate of omission of axillary node dissection in case of micrometastasis increased (Bilimoria) despite any strong proof has been demonstrated.

The omission of axillary node dissection in case of positive sentinel node may have strong practical impacts on patients but also on medical and economical aspects: in avoiding a prolonged hospitalisation, secondary morbidities due to axillary dissection requiring secondary care and their costs, as well as costs for secondary axillary dissection (14 to 25% in case of positive sentinel node) and finally shortening surgery duration.

The main investigator propose a Non Inferiority Randomized Multicenter Phase III Trial of Axillary Node Dissection Versus no Axillary Node Dissection in Case of Positive Sentinel Lymph Node in Invasive Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. - Patient aged 18 years and above,
2. - Patient with invasive breast cancer histologically proven or cytologically proven by fine needle biopsy,
3. - Patient with a unifocal tumor T0 - T1 - T2 up to 5 cm (clinical or in imagery), without previous therapy (neoadjuvant chemotherapy or hormone therapy),
4. - Patient with clinical N0 status,
5. - Absence of clinically detectable metastases known,

6- Patients for whom conservative surgery with sentinel lymph node (SLN) technique is feasible from the start in terms of carcinologic,

7 -All patients with lymph node involvement (GS+), whatever the size of the metastasis (macro-metastasis, micro-metastasis, cellular cluster or isolated tumor cells),

8 - Patient affiliated to a social security system or benefiting from such a system,

9 - Signed consent to participate.

Exclusion Criteria:

1. - Tumor of more than 5 cm
2. - Indication of neoadjuvant therapy by chemotherapy or hormone therapy
3. - History of breast cancer (ipsilateral, ie recurrence, or contralateral breast)
4. - History of any other invasive cancer other than a past cutaneous cancer correctly treated
5. - Initial metastatic disease known
6. - Presence of clinical axillary adenopathy
7. - Contra-indication to surgical excision
8. - Contra-indication to the SLN technique
9. - Pregnant women, of child-bearing potential, or lactating women

10- Patient deprived of liberty or under supervision of a guardian

11- Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2228 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Disease Free survival | Time to relapse or progression up to 10 years
  time from randomization to relapse or death.

SECONDARY OUTCOMES:
axillary recurrence rate | Time to local relapse up to 10 years
  Estimate the incidence of axillary recurrence after surgery followed by axillary dissection or after surgery alone.
Overall survival | Time to death up to 10 years
  Time from randomization to date of death

CONTACTS AND LOCATIONS:
Overall Officials: Gilles HOUVENAEGHEL, MD, PHD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Gilles HOUVENAEGHEL, PHD, Marseille, France

REFERENCES:
- [Background] Giuliano AE, Ballman KV, McCall L, Beitsch PD, Brennan MB, Kelemen PR, Ollila DW, Hansen NM, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Morrow M. Effect of Axillary Dissection vs No Axillary Dissection on 10-Year Overall Survival Among Women With Invasive Breast Cancer and Sentinel Node Metastasis: The ACOSOG Z0011 (Alliance) Randomized Clinical Trial. JAMA. 2017 Sep 12;318(10):918-926. doi: 10.1001/jama.2017.11470. PMID 28898379
- [Background] Donker M, van Tienhoven G, Straver ME, Meijnen P, van de Velde CJ, Mansel RE, Cataliotti L, Westenberg AH, Klinkenbijl JH, Orzalesi L, Bouma WH, van der Mijle HC, Nieuwenhuijzen GA, Veltkamp SC, Slaets L, Duez NJ, de Graaf PW, van Dalen T, Marinelli A, Rijna H, Snoj M, Bundred NJ, Merkus JW, Belkacemi Y, Petignat P, Schinagl DA, Coens C, Messina CG, Bogaerts J, Rutgers EJ. Radiotherapy or surgery of the axilla after a positive sentinel node in breast cancer (EORTC 10981-22023 AMAROS): a randomised, multicentre, open-label, phase 3 non-inferiority trial. Lancet Oncol. 2014 Nov;15(12):1303-10. doi: 10.1016/S1470-2045(14)70460-7. Epub 2014 Oct 15. PMID 25439688
- [Background] Jagsi R, Chadha M, Moni J, Ballman K, Laurie F, Buchholz TA, Giuliano A, Haffty BG. Radiation field design in the ACOSOG Z0011 (Alliance) Trial. J Clin Oncol. 2014 Nov 10;32(32):3600-6. doi: 10.1200/JCO.2014.56.5838. Epub 2014 Aug 18. PMID 25135994
- [Result] Houvenaeghel G, Cohen M, Raro P, De Troyer J, de Lara CT, Gimbergues P, Gauthier T, Faure-Virelizier C, Vaini-Cowen V, Lantheaume S, Regis C, Darai E, Ceccato V, D'Halluin G, Del Piano F, Villet R, Jouve E, Beedassy B, Theret P, Gabelle P, Zinzindohoue C, Opinel P, Marsollier-Ferrer C, Dhainaut-Speyer C, Colombo PE, Lambaudie E, Tallet A, Boher JM; Others investigators (SERC trial group). Overview of the pathological results and treatment characteristics in the first 1000 patients randomized in the SERC trial: axillary dissection versus no axillary dissection in patients with involved sentinel node. BMC Cancer. 2018 Nov 21;18(1):1153. doi: 10.1186/s12885-018-5053-7. PMID 30463611
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr